CLINICAL TRIAL: NCT07275970
Title: An Open-Label, Phase 1 Study of the Safety Pharmacokinetic Profile, and Preliminary Efficacy, of Organic Whole Psilocybin-Containing Mushrooms in Patients Suffering From PTSD
Brief Title: Safety and Preliminary Efficacy of Organic Whole Psilocybin-Containing Mushrooms to Treat Patients Suffering From PTSD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sue Sisley (Other)
Collaborators: Scottsdale Research Institute (Other)
Responsible Party: Sponsor-Investigator, Sue Sisley, Principal Investigator, Scottsdale Research Institute
Organization: Scottsdale Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRI-HRTT21
Record Dates: First submitted 2025-11-26; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: PTSD
Keywords: ptsd; psilocybin
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Hallucinogens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 30mg of psilocybin administered orally in a single dosing session (Experimental)
  Interventions: Drug: Psychedelic

INTERVENTIONS:
Drug: Psychedelic — Organic Whole Psilocybin-Containing Mushrooms

SUMMARY:
This study will examine the safety and preliminary efficacy of psilocybin mushrooms to treat adults with PTSD. Up to 24 participants will take part in this study. Each participant will ingest psilocybin from dried mushrooms in a chocolate formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals ≥ 18 years of age
2. Have a diagnosis of Post-Traumatic Stress Disorder (PTSD) as defined:

   * Meet Diagnostic and Statistical Manual-5th edition (DSM-5) criteria for current PTSD with a duration of 6 months or longer as assessed by a study psychiatrist.
   * Determination of at least one traumatic event as determined by the LEC-5
   * A score of at least 33 on the PCL-5
3. Willing and able to provide signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

   •Willingly agreed to provide verbal consent to provide needed pre-screening information, including medical history, concomitant medications, etc., prior to signing the ICF.
4. Be willing to commit to self-administering the study drug, to completing the QoL and PRO instruments, and attending all study visits.
5. Participants must be able to evaluate their average pain on the BPI (Brief Pain Inventory) over the past week.
6. Acceptable renal functioning as determined by no significant prior medical history and results of clinical laboratory evaluations done at Screening and on Day 1 (e.g., eGFR >45 (mL/min/1.73 m2))
7. Acceptable hepatic functioning as determined by no significant prior medical history and results of clinical laboratory evaluations done at Screening and on Day 1 (e.g., liver enzymes ≤1.5x the upper limit of normal, 'ULN')
8. Agree to only use the psilocybin mushroom provided by site staff and not use any other psilocybin (or similar drug) in any form for at least 30 days prior to Study Day 1 and for 30 days following the single-dose study drug treatment.
9. Is willing to wear, sync daily, and charge twice weekly a provisioned health tracking wearable device every day during sleep and daily activity. If the participant already has the same, or compatible device, they can use their own.
10. Agree to not use any psychoactive drugs, partake alcoholic beverages, self-administer ondansetron (or other selective serotonin reuptake inhibitors 'SSRIs', serotonin-norepinephrine reuptake inhibitors, 'SNRIs' and monoamine oxidase inhibits, 'MAOs'), cannabis, and/or any other non-routine PRN medications within 24 hours of Study Day 1. Exceptions include daily use of caffeine, nicotine, and opioid pain medication
11. Be stable on any pre-study medications and/or psychotherapy regimen prior to study entry. Agree to inform physician(s)/clinician(s) providing current care about your participation in the study (or permit the research site study staff to do so). Agree to report any changes in medication or psychotherapy treatment regimen during the study, to study staff.
12. If female and of childbearing potential, the participant is eligible for the trial only with a negative urine pregnancy test during Screening and on Study Day 1. [If a result is uncertain (e.g., potential false positive), a serum human chorionic gonadotropin (hHCG) test may be performed prior to the administration of the study drug.] Fertile females agree to use a highly effective form of birth control during the 30-day posttreatment period and must confirm that they have no intent to try to become pregnant or any need to breastfeed during this period.

    • Adequate birth control methods include intrauterine device (IUD), injected or implanted hormonal methods, oral hormones plus a barrier contraception, or double barrier contraception. Two forms of contraception are required with any barrier method or oral hormones (i.e., condom and diaphragm, condom or diaphragm and spermicide, oral hormonal contraceptives and spermicide or condom). Not of childbearing potential is defined as permanent sterilization or postmenopausal females.
13. Be proficient in reading and writing in English and able to effectively communicate with site staff.
14. Agree not to participate in any other interventional clinical trials during the study.

Exclusion Criteria:

1. Currently uncontrolled hypertension. (>140/90 at Screening and >145/95 on Study Day 1).
2. History of recent seizure (within 3 months of Study Day 1).
3. History of stroke or transient ischemic attacks.
4. Preexisting history of valvulopathy or pulmonary hypertension.
5. A marked prolongation of QT interval (i.e., QT ≥450 msec) over a series of 3 ECGs performed within 5-6 minutes.

Currently uncontrolled diabetes (HbA1c > 8.0%). 7. Potential for adverse drug-drug interactions such as the use of centrally-acting serotonergic agents within 24 hours prior to and for 72 hours following study drug administration on Study Day 1.

8. Significant suicide risk defined by (1) suicidal ideation as endorsed on items 4 or 5 on the Columbia Suicidal Severity Rating Scale (C-SSRS) within the last 6 months, at Screening, or at Baseline (Visit 1), or; (2) suicidal behaviors within the last 12 months as assessed by C-SSRS.

9. Patients with severe anxiety and depression measured as following: Participants with scores of 15 & above on Generalized Anxiety Disorder-7 (GAD-7) scale, and/or with scores of 20 & above on Patient Health Questionnaire-9 (PHQ -9).

10. Are pregnant or nursing or are women of childbearing potential who are not practicing a highly effective means of birth control.

11. Have any allergies or contraindication to psilocybin mushrooms. 12. Current users of psilocybin, LSD, DMT, Ayahuasca, Peyote, mescaline, and ketamine over the past 30 days will not qualify for the study unless the use of these agents is stopped for 30 days prior to Study Day 1 and the participant agrees to not use these (or similar) agents for 30 days after Study Day 1.

13. Are not able to attend face-to-face visits at the study site or plan to move out of the area prior to the 3-month LTFU visit.

14. Have any current problem that, in the opinion of the Investigator or Medical Monitor, might interfere with an individual's participation in the study or confound the assessment of safety and/or efficacy of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number/Incidence of adverse events (AEs), and serious adverse events (SAEs) graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. | From dosing to 3-month follow-up
Number/Incidence of Mental and Psychotic AE's | From dosing to 3-month follow-up

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Psilocin | pre-dose to 8-hours post-dose
  Cmax will be determined using non-compartmental analysis of plasma psilocin concentrations.
Time to Maximum Plasma Concentration (Tmax) of Psilocin | Pre-dose to 8 hours post-dose
  Tmax will be calculated as the time point at which the maximum psilocin concentration occurs.
Area Under the Curve (AUC₀-₈) for Psilocin | Pre-dose to 8 hours post-dose
  AUC₀-₈ will be calculated using the linear trapezoidal method to assess total psilocin exposure.

CONTACTS AND LOCATIONS:
Locations (1):
- Scottsdale Research Institute, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided